CLINICAL TRIAL: NCT06726031
Title: The Effect of Using Virtual Reality Glasses on Anxiety-related Radial Vasospasm in Patients Undergoing Transradial Coronary Angiography
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Ahmet Burak KECECİ, researcher doctor, Mersin University
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MersinU-CAR-ABK-01
Record Dates: First submitted 2024-11-29; First posted 2024-12-10 (Actual); Last update posted 2024-12-10 (Actual); Status verified 2024-12

CONDITIONS: Radial Artery Spasm; Radial Artery Access; Virtual Reality
Keywords: radial artery spasm; virtual reality; anxiety
MeSH Terms: conditions — Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- control group (No Intervention): Participants in this group will not undergo VR glasses application during transradial coronary angiography.
- VR Glass Group (Active Comparator): Participants in this group will use VR glasses during transradial coronary angiography. With the help of VR glasses, patients will be shown visuals based on nature and listen to calming sounds.
  Interventions: Device: wearing VR glass

INTERVENTIONS:
Device: wearing VR glass — The intervention is the application of VR headsets during the procedure for patients who were previously indicated for transradial coronary angiography and were randomized to the VR headset group.
  Arms: VR Glass Group

SUMMARY:
Compared to transfemoral access, transradial access is a safe and effective method for coronary interventions, associated with lower rates of vascular complications, including major bleeding. Additionally, it facilitates early ambulation and reduces post-procedural hospital stays. As a result, current guidelines now recommend transradial access as the preferred approach for coronary interventional procedures. However, the most commonly recognized limitation of this method is radial artery spasm (RAS).

The radial artery is more susceptible to spasm than other peripheral arteries due to its thicker muscular layer and the predominance of alpha-adrenergic receptors. RAS can sometimes limit the advantages of transradial access, prolong procedural duration, or even lead to procedural failure and termination. Consequently, the prevention of potential causes of RAS has garnered significant interest.

The reported incidence of RAS ranges between 7.8% and 25%. These rates are notably high for diagnostic procedures, underscoring the importance of identifying and addressing risk factors before the intervention. The literature identifies several risk factors for RAS, including female sex, advanced age, smaller radial artery diameter, and the number of interventions performed.

Cardiac procedures frequently induce pain and anxiety in patients. The prevalence of anxiety disorders among patients with cardiovascular diseases can reach up to 15%, with cardiac procedures exacerbating these conditions, resulting in anxiety prevalence rates as high as 72%.

Given the limitations of pharmacological approaches in managing pain and anxiety, innovative digital solutions such as virtual reality (VR) have been proposed. However, VR was not found to have a statistically significant effect on pain levels.

The literature review revealed that, based on the current understanding, no prior studies have investigated the impact of VR headset use on anxiety-induced vasospasm in patients undergoing transradial coronary angiography. Therefore, the study aimed to explore whether VR applications could influence the successful completion of this widely performed procedure worldwide.

ELIGIBILITY:
Inclusion Criteria:

* Indicated for coronary angiography via the transradial approach for reasons other than Acute Coronary Syndrome.
* Patients with no prior history of coronary angiography
* Patients aged 18 years and older
* Patients who are conscious, oriented, cooperative, and able to read and understand Turkish.
* Patients without any physical issues that would prevent the use of virtual reality glasses.
* Patients with no known malignancy, neuropsychiatric disorders, or diagnosed anxiety disorders.
* Patients who agree to participate in the study and sign the "Informed Consent Form" will be included.

Exclusion Criteria:

* Patients indicated for coronary angiography due to Acute Coronary Syndrome,
* Patients undergoing coronary angiography via an approach other than the transradial route,
* Patients under the age of 18,
* Patients who are unconscious, disoriented, or uncooperative,
* Patients who cannot read or understand Turkish,
* Patients with physical issues preventing the use of virtual reality glasses,
* Patients with known neuropsychiatric disorders, diagnosed anxiety disorders, or those receiving antidepressant or anxiolytic treatment,
* Patients with malignancy,
* Patients who do not agree to participate or who do not sign the "Informed Consent Form" will be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
the Visual Analog Scale (VAS) | day 1
  Visual Analog Scale (VAS) is used to convert certain non-quantifiable values into numerical data. A 100-mm line is marked with two extreme descriptions of the parameter being evaluated at each end. Patients are asked to indicate their current state on the line by drawing a mark, placing a dot, or pointing to a specific location.
  For example, in the case of pain, one end of the line might read "no pain at all," and the other end "worst imaginable pain." The patient marks the point on the line that best represents their current pain level. The distance from the "no pain" end to the point marked by the patient represents the intensity of the pain they are experiencing.
  The length of the line between these two points serves as a measure of the patient's subjective experience.

SECONDARY OUTCOMES:
the State-Trait Anxiety Inventory (STAI) | day 1
  The STAI (State-Trait Anxiety Inventory) is a psychological tool developed to assess individuals' anxiety levels and consists of a total of 40 questions. The scale addresses anxiety in two distinct dimensions: State Anxiety and Trait Anxiety. State anxiety measures the individual's temporary level of anxiety in response to a specific and transient situation, while trait anxiety evaluates the individual's general tendency to experience anxiety and their predisposition to perceive anxiety as a personality trait. Both subscales consist of 20 questions, and individuals are asked to indicate how much the given statements apply to them.

CONTACTS AND LOCATIONS:
Overall Officials: ahmet b KECECI, Research Assistant, Principal Investigator — Mersin University faculty of medicine
Locations (1):
- Mersin University Faculty of Medicine, Mersin, Yenisehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided